CLINICAL TRIAL: NCT04652180
Title: Clinical Trial Of Safety Of Robot-assisted Thoracic Approach Verus Open Transthoracic Esophagectomy in Esophageal Cancer.
Brief Title: Robot-assisted Thoracic Approach Versus Open Transthoracic Esophagectomy .
Acronym: CIR·ROB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: University of Barcelona (Other)
Responsible Party: Principal Investigator, Carla Bettonica, PhD, PhD. Department of Esophagogastric Surgery, Hospital Universitari de Bellvitge, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUB-CIR-ROB-2020-01
Record Dates: First submitted 2020-11-09; First posted 2020-12-03 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Esophageal Cancer; Esophageal Carcinoma; Postoperative Complications
MeSH Terms: conditions — Esophageal Neoplasms; Postoperative Complications | interventions — Esophagectomy

STUDY DESIGN:
Intervention Model Description: Monocentre randomized controlled parallel-group, phase IV, superiority trial. The main purpose is to demonstrate the superiority of robot-assisted thoracic approach over thoracotomy (conventional surgery) in decreasing respiratory and overall complications in Ivor Lewis-type esophagectomy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robot-assisted thoracic approach in Ivor Lewis esophagectomy (Experimental): Robot-assisted thoracic approach in Ivor Lewis esophagectomy with gastric conduit formation. Abdominal approach will be performed by laparoscopy.
  Interventions: Procedure: Esophagectomy
- Open transthoracic approach in Ivor Lewis esophagectomy (Active Comparator): Traditional open transthoracic esophagectomy with gastric conduit formation. Abdominal approach will be performed by laparoscopy.
  Interventions: Procedure: Esophagectomy

INTERVENTIONS:
Procedure: Esophagectomy — In this monocentre randomized controlled trial, we compare robot-assisted thoracic approach with conventional open transthoracic Ivor Lewis esophagectomy.
  Other Names: Robot-assisted minimally invasive esophagectomy; Robot-assisted thoracic approach in Ivor Lewis esophagectomy

SUMMARY:
This is a randomized controlled trial designed to compare robot-assisted thoracic approach with open transthoracic esophagectomy (Ivor Lewis technique) as a surgical treatment for resectable esophageal cancer.

If our hypothesis is proved correct, robot-assisted thoracic approach will result in a lower percentage of respiratory and overall postoperative complications, lower blood loss, shorter hospital stay, but with at least similar oncologic outcomes and better postoperative quality of life compared with the open transthoracic esophagectomy (current standard).

DETAILED DESCRIPTION:
Rationale: Esophageal cancer represents the fifth most common tumor of cancers of the digestive system in Spain, between the ten most common cancers and the sixth leading cause of cancer death in the world. Among the standard modalities for treatment with curative intention, surgery is available, in combination with neoadjuvant (pre-surgery) and/or adjuvant (post-surgery) chemotherapy and radiation therapy. Esophageal surgery is crucial to improve overall survival in patients with esophageal cancer.

Surgical treatment is based on esophageal resection and reconstruction of digestive transit, as well as a correct lymphadenectomy. One of the techniques used is Ivor Lewis transthoracic esophagectomy. Classically, thoracic approach has been done by open approach (thoracotomy), with minimally invasive (laparoscopy) abdominal approach, a reality in our centre and in most European centres.

Postoperative comorbidity, specially respiratory complications, occur approximately in half of patients with esophagectomy with thoracotomy (open approach). Although current clinical trials have reported advantages over minimally invasive esophagectomy (MI), at the time, most esophageal surgery is performed by open approach. More studies are needed to clarify the role of minimally invasive esophagectomy in esophageal cancer, so as to provide evidence about the comorbidity and effectiveness of surgical robot-assisted technique.

If our hypothesis is proved correct, robot-assisted thoracic approach will result in a lower percentage of respiratory and overall postoperative complications, lower blood loss, shorter hospital stay, but with at least similar oncologic outcomes and better postoperative quality of life compared with the open transthoracic esophagectomy (current standard).

Objective: Evaluate the benefits, risks and cost-efficiency of Robot-assisted thoracic approach as a better approach to open transthoracic Ivor Lewis esophagectomy as treatment for esophageal cancer.

Study design: This is an investigator-initiated and investigator-driven monocentre randomized controlled parallel-group, phase IV, superiority trial.

Study populations: Patients (age ≥ 18) with histologically proven surgical resectable (cT1-4a, N0-3, M0) adenocarcinoma, squamous cell carcinoma, undifferentiated esophageal carcinoma or carcinomas of the esophagogastric junction (EGJ) (Siewert I or II) candidate to Ivor Lewis Esophagectomy.

Intervention:108 patients will be randomly allocated to either A) Robot-assisted thoracic approach or B) Open transthoracic esophagectomy, in Ivor Lewis technique. In both groups the abdominal approach will be performed by laparoscopy (minimally invasive).

Patients will receive the following interventions:

Group A. Robot-assisted thoracic approach in Ivor Lewis esophagectomy. Group B. Open transthoracic approach (thoracotomy) in Ivor Lewis esophagectomy.

Both surgical techniques are used in our usual clinical practice of the General and Digestive Surgery Department of the Bellvitge University Hospital (HUB).

Main study parameters/endpoints: Primary outcome is the percentage of respiratory and overall complications as stated by the modified Clavien-Dindo classification (MCDC).

Secondary outcomes are individual components of the primary endpoint (major and minor complications), (in hospital) mortality, R0 resections, oncologic outcomes, postoperative recovery, cost-effectiveness and quality of life.

Follow-up:84±3 days after hospital discharge.

NOTE: The project consists of a clinical trial and an extension study to assess the free-survival of 3 and 5 years from surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Histologically proven adenocarcinoma, squamous cell carcinoma, undifferentiated carcinoma or carcinoma of the gastro-esophageal junction (GEJ) Siewert I or II.
* Surgical resectable (T1-4a, N0-3, M0).
* Childbearing potential women (period between menarche and menopause), pregnancy negative test is mandatory.
* Written informed consent.

Exclusion Criteria:

* Stage IV or GEJ Siewert III esophageal cancer.
* Contraindication of transthoracic esophagectomy in two fields.
* Pre- or concomitant cancer or conditions which interferes with the study (e.g. prior thoracic surgery or trauma. Rationale: these patients may undergo open resection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2020-11-06 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Respiratory postoperative complications. | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks up to 84+/-3 days from hospital discharge.
  The primary outcome of this study is the percentage of respiratory complications as stated by the modified Clavien-Dindo classification of surgical complications (MCDC).
  by means of AME chest approach by robot and thoracotomy (classic surgery).

SECONDARY OUTCOMES:
Postoperative complications. | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks up to 84+/-3 days from hospital discharge.
  Estimate the percentage of overall complications as stated by the modified Clavien-Dindo classification of surgical complications (MCDC) by means of Robot-assisted thoracic approach and thoracotomy (classic surgery).
Individual components of the primary endpoint (major and minor complications). | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks up to 84+/-3 days from hospital discharge
  Major complications (MCDC Grade 2-4): anastomotic leakage (clinical or radiologic diagnosis), anastomotic stenosis, chylothorax (chylous leakage, presence of chylous in chest tubes or indication start medium chain triglycerides containing tube feeding), gastric tube necrosis (proven by gastroscopy), pulmonary embolus, pneumothorax, deep vein thrombosis, myocardial infarction, vocal cord palsy or paralysis.
  Minor complications (MCDC Grade 1): wound infections, pleural effusions, delayed gastric emptying.
  All these postoperative complications will be properly and separately recorded in the electronic collection database.
Postoperative mortality (during hospital stay up to 84+/-3 days after discharge). | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks up to 84+/-3 days from hospital discharge.
  (In hospital) mortality and mortality within 14+/-2 days and 84+/-3 days after hospital discharge will be reported. The cause of death will be noted.
Operation related events. | Day of surgery, up to 24 hours after surgery.
  Operation time is defined as time from incision until closure (minutes) for both the thoracic and the abdominal phase of the procedure. For the robotic approach, set up time will be recorded separately. Unexpected events and complications occuring during operation will be recorded (e.g. massive hemorrhage, perforation of other organs). Blood loss during operation (ml, per phase). In case of conversion to thoracotomy or laparotomy the reason for conversion has tp be explained (absolute numbers/percentage).
Postoperative recovery. | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.
  Pain: type and dose of used analgesics will be noted during the hospital admission period and noted during the follow-up period. Unit of measure: Visual Analog Score for pain.
  Length of intensive care unit (ICU) (days). Length of hospital stay (days).
R0 resections (%). | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks and 14+/- days after discharge.
  The pathological analysis will be finished within 2-3 weeks after surgery.
Oncologic outcomes. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 84+/-3 days after discharge.
  Overall survival within the first 84+/-3 days. NOTE: 2, 3 and 5 year disease free and overall survival will be reported in the study of extension .
Postoperative quality of life. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 84+/-3 days after discharge.
  Postoperative quality of life will be assessed through Physicians Global Assessment to measure quality of life:
  Questionnaires EORTC QLQ-C30 and EQ-5D will be required from 14+/-2 up to 84+/-3 days after hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Leandre Farran, PhD Surgeon, Study Director
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately following publication and ending 11 months after publication.
Access Criteria: Researches who wish to access the data with a methodological proposal. Types of analyses: to achieve aims in the approved proposal. Mechanism:Proposals should be directed to nataliacornellagcirurgia@gmail.com. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Result] Stahl M, Mariette C, Haustermans K, Cervantes A, Arnold D; ESMO Guidelines Working Group. Oesophageal cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2013 Oct;24 Suppl 6:vi51-6. doi: 10.1093/annonc/mdt342. No abstract available. PMID 24078662
- [Result] Inderhees S, Dubecz A. [Hybrid minimally invasive esophagectomy for esophageal cancer-MIRO trial]. Chirurg. 2019 Aug;90(8):677. doi: 10.1007/s00104-019-0983-4. No abstract available. German. PMID 31127335
- [Result] van der Sluis PC, van der Horst S, May AM, Schippers C, Brosens LAA, Joore HCA, Kroese CC, Haj Mohammad N, Mook S, Vleggaar FP, Borel Rinkes IHM, Ruurda JP, van Hillegersberg R. Robot-assisted Minimally Invasive Thoracolaparoscopic Esophagectomy Versus Open Transthoracic Esophagectomy for Resectable Esophageal Cancer: A Randomized Controlled Trial. Ann Surg. 2019 Apr;269(4):621-630. doi: 10.1097/SLA.0000000000003031. PMID 30308612
- [Result] Straatman J, van der Wielen N, Cuesta MA, Daams F, Roig Garcia J, Bonavina L, Rosman C, van Berge Henegouwen MI, Gisbertz SS, van der Peet DL. Minimally Invasive Versus Open Esophageal Resection: Three-year Follow-up of the Previously Reported Randomized Controlled Trial: the TIME Trial. Ann Surg. 2017 Aug;266(2):232-236. doi: 10.1097/SLA.0000000000002171. PMID 28187044
- [Result] Avery KN, Metcalfe C, Berrisford R, Barham CP, Donovan JL, Elliott J, Falk SJ, Goldin R, Hanna G, Hollowood AA, Krysztopik R, Noble S, Sanders G, Streets CG, Titcomb DR, Wheatley T, Blazeby JM. The feasibility of a randomized controlled trial of esophagectomy for esophageal cancer--the ROMIO (Randomized Oesophagectomy: Minimally Invasive or Open) study: protocol for a randomized controlled trial. Trials. 2014 Jun 2;15:200. doi: 10.1186/1745-6215-15-200. PMID 24888266
- [Result] Brierley RC, Gaunt D, Metcalfe C, Blazeby JM, Blencowe NS, Jepson M, Berrisford RG, Avery KNL, Hollingworth W, Rice CT, Moure-Fernandez A, Wong N, Nicklin J, Skilton A, Boddy A, Byrne JP, Underwood T, Vohra R, Catton JA, Pursnani K, Melhado R, Alkhaffaf B, Krysztopik R, Lamb P, Culliford L, Rogers C, Howes B, Chalmers K, Cousins S, Elliott J, Donovan J, Heys R, Wickens RA, Wilkerson P, Hollowood A, Streets C, Titcomb D, Humphreys ML, Wheatley T, Sanders G, Ariyarathenam A, Kelly J, Noble F, Couper G, Skipworth RJE, Deans C, Ubhi S, Williams R, Bowrey D, Exon D, Turner P, Daya Shetty V, Chaparala R, Akhtar K, Farooq N, Parsons SL, Welch NT, Houlihan RJ, Smith J, Schranz R, Rea N, Cooke J, Williams A, Hindmarsh C, Maitland S, Howie L, Barham CP. Laparoscopically assisted versus open oesophagectomy for patients with oesophageal cancer-the Randomised Oesophagectomy: Minimally Invasive or Open (ROMIO) study: protocol for a randomised controlled trial (RCT). BMJ Open. 2019 Nov 19;9(11):e030907. doi: 10.1136/bmjopen-2019-030907. PMID 31748296
- [Result] Luketich JD, Pennathur A, Awais O, Levy RM, Keeley S, Shende M, Christie NA, Weksler B, Landreneau RJ, Abbas G, Schuchert MJ, Nason KS. Outcomes after minimally invasive esophagectomy: review of over 1000 patients. Ann Surg. 2012 Jul;256(1):95-103. doi: 10.1097/SLA.0b013e3182590603. PMID 22668811
- [Result] Pennathur A, Luketich JD, Landreneau RJ, Ward J, Christie NA, Gibson MK, Schuchert M, Cooper K, Land SR, Belani CP. Long-term results of a phase II trial of neoadjuvant chemotherapy followed by esophagectomy for locally advanced esophageal neoplasm. Ann Thorac Surg. 2008 Jun;85(6):1930-6; discussion 1936-7. doi: 10.1016/j.athoracsur.2008.01.097. PMID 18498797
- See also: Esophageal cancer — http://seom.org
- See also: Survival — http://seer.cancer.gov
- See also: Cancer Staging — http://cancerstaging.org
- See also: Diagnosis — http://www.cancer.org

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT04652180/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT04652180/ICF_001.pdf